CLINICAL TRIAL: NCT03219268
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation Study of MGD013, A Bispecific DART® Protein Binding PD-1 and LAG-3 in Patients With Unresectable or Metastatic Neoplasms
Brief Title: A Study of MGD013 in Patients With Unresectable or Metastatic Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD013-01
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumors; Hematologic Neoplasms; Ovarian Cancer; HER2-positive Advanced Solid Tumors; Non Small Cell Lung Cancer; Small-cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Cholangiocarcinoma; Cervical Cancer; TNBC - Triple-Negative Breast Cancer
MeSH Terms: conditions — Hematologic Neoplasms; Ovarian Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Cholangiocarcinoma; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms | interventions — margetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Tebotelimab: 1 mg (Experimental)
  Interventions: Biological: tebotelimab 1 mg
- Tebotelimab 3 mg (Experimental)
  Interventions: Biological: tebotelimab 3 mg
- Tebotelimab: 10 mg (Experimental)
  Interventions: Biological: tebotelimab 10 mg
- Tebotelimab: 30 mg (Experimental)
  Interventions: Biological: tebotelimab 30 mg
- Tebotelimab: 120 mg (Experimental)
  Interventions: Biological: tebotelimab 120 mg
- Tebotelimab: 400 mg (Experimental)
  Interventions: Biological: tebotelimab 400 mg
- Tebotelimab: 600 mg (Experimental)
  Interventions: Biological: tebotelimab 600 mg
- Tebotelimab: 800 mg (Experimental)
  Interventions: Biological: tebotelimab 800 mg
- Tebotelimab: 1200 mg (Experimental)
  Interventions: Biological: tebotelimab 1200 mg
- Combination cohort 1 (Experimental): Tebotelimab and margetuximab
  Interventions: Biological: tebotelimab 300 mg; Biological: margetuximab
- Combination Cohort 2 (Experimental): Tebotelimab and margetuximab
  Interventions: Biological: tebotelimab 600 mg; Biological: margetuximab
- Monotherapy Cohort Expansion (Experimental): Monotherapy expansion at 600 mg
  Interventions: Biological: tebotelimab 600 mg

INTERVENTIONS:
Biological: tebotelimab 1 mg — 1 mg IV every other week
  Other Names: MGD013
  Arms: Tebotelimab: 1 mg
Biological: tebotelimab 3 mg — 3 mg IV every other week
  Other Names: MGD013
  Arms: Tebotelimab 3 mg
Biological: tebotelimab 10 mg — 10 mg IV every other week
  Other Names: MGD013
  Arms: Tebotelimab: 10 mg
Biological: tebotelimab 30 mg — 30 mg IV every other week
  Other Names: MGD013
  Arms: Tebotelimab: 30 mg
Biological: tebotelimab 120 mg — 120 mg IV every other week
  Other Names: MGD013
  Arms: Tebotelimab: 120 mg
Biological: tebotelimab 300 mg — 300 mg IV every other wee
  Other Names: MGD013
  Arms: Combination cohort 1
Biological: tebotelimab 400 mg — 400 mg IV every other wee
  Other Names: MGD013
  Arms: Tebotelimab: 400 mg
Biological: tebotelimab 600 mg — 600 mg IV every other week
  Other Names: MGD013
  Arms: Combination Cohort 2; Monotherapy Cohort Expansion; Tebotelimab: 600 mg
Biological: tebotelimab 800 mg — 800 mg IV every other week
  Other Names: MGD013
  Arms: Tebotelimab: 800 mg
Biological: tebotelimab 1200 mg — 1200 mg IV every other week
  Other Names: MGD013
  Arms: Tebotelimab: 1200 mg
Biological: margetuximab — 15 mg/kg IV every 3 weeks
  Other Names: MGAH22; Margenza
  Arms: Combination Cohort 2; Combination cohort 1

SUMMARY:
The primary goal of this Phase 1 study is to characterize the safety and tolerability of tebotelimab and establish the maximum tolerated dose (MTD) of tebotelimab in advanced solid tumors, and tebotelimab in combination with margetuximab in HER2+ advanced solid tumors. Pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD), and the anti-tumor activity of tebotelimab will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, locally advanced unresectable or metastatic solid tumors (or hematologic malignancies, Cohort Expansion only) for whom no approved therapy with demonstrated clinical benefit is available or standard treatment was declined.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy ≥ 12 weeks
* Measurable disease
* Tissue specimen available for retrospective analysis of PD-1, PD-L1, LAG-3, and MHC-II expression
* Acceptable laboratory parameters

HER2+ Cohort:

- Locally advanced or metastatic HER2+ locally advanced or metastatic solid tumors, regardless of organ of origin.

i. The cancer must have progressed following standard therapy, or has progressed during or after HER2-directed therapy if approved and available for patients with HER2+ breast, gastric, or gastroesophageal junction cancer.

ii. History of HER2 positivity defined as 3+ by IHC or 2+ by Immunohistochemistry (IHC) in combination with in situ hybridization (ISH) positivity most recent tumor biopsy.

* All patients in the HER2+ cohort must be willing to provide consent for a baseline and on-treatment tumor biopsy during the screening period and within 14 days prior to Cycle 3 Day 1. Exceptions may be made based on a medical contraindication at the discretion of the Sponsor's Medical Monitor. This requirement will be discontinued after an adequate number of samples are collected, as determined by the Sponsor.

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases or primary CNS lymphoma
* History of allogeneic bone marrow, stem-cell, or solid organ transplant
* History of known or suspected autoimmune disease with the specific exceptions of vitiligo, resolved childhood atopic dermatitis, psoriasis not requiring systemic treatment (within the past 2 years), and patients with a history of Grave's disease that are now euthyroid clinically and by laboratory testing.
* Treatment with any systemic chemotherapy within 3 weeks prior to the initiation of study drug; treatment with biologics or investigational therapy within the 4 weeks prior to the initiation of study drug.
* Major surgery within 4 weeks prior to the initiation of study drug.
* Prior treatment with combination of monoclonal antibodies against PD-1 and LAG-3 (Cohort Expansion only).
* Treatment with radiation therapy within 2 weeks prior to the initiation of study drug.
* Clinically significant cardiovascular disease.
* QTcF prolongation > 480 milliseconds
* HER2+ cohort: left ventricular ejection fraction less than 50%
* Clinically significant pulmonary compromise, including a requirement for supplemental oxygen use to maintain adequate oxygenation.
* Active pneumonitis or history of non-infectious pneumonitis.
* Clinically significant gastrointestinal disorders.
* Evidence of active viral, bacterial, or systemic fungal infection requiring parenteral treatment within 7 days prior to the initiation of study drug.
* Known history of positive testing for human immunodeficiency virus or history of acquired immune deficiency syndrome.
* Known history of hepatitis B (except in hepatocellular carcinoma) or hepatitis C infection or known positive test for hepatitis B surface antigen, hepatitis B core antigen, or hepatitis C polymerase chain reaction (PCR)
* Vaccination with any live virus vaccine within 4 weeks prior to the initiation of study drug administration. Inactivated annual influenza vaccination is allowed
* Dementia or altered mental status that would preclude understanding and rendering of informed consent
* Confirmed or presumed COVID-19/SARS-CoV-2 infection. While SARS-CoV-2 testing is not mandatory for study entry, testing should follow local clinical practice guidelines/standards. Patients with a positive test result for SARS-CoV-2 infection, known asymptomatic infection, or presumed infection are excluded. Patients may be considered eligible after a resolved SARS-CoV-2 infection once he or she remains afebrile for at least 72 hours and after other SARS-CoV-2-related symptoms have fully recovered to baseline for a minimum of 72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events (TEAE) as assessed by CTCAE v4.03 (tebotelimab monotherapy) | up to 24 months
  Safety
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit.
Number of participants with Treatment-Emergent Adverse Events as assessed by CTCAE v4.03 (tebotelimab plus margetuximab) | up to 24 months
  Safety

SECONDARY OUTCOMES:
Area Under the Plasma Concentration versus Time Curve (AUC) of tebotelimab | From Day 1 to Day 15 after the first and second doses
  AUC
Maximum Plasma Concentration (Cmax) of tebotelimab and tebotelimab plus margetuximab | At the end of infusion on Study Days 1, 15, 29 and 43 in Cycles 1 and 2 and on Study Day 1 for all subsequent cycles until treatment discontinuation, up to 2 years
  Cmax
Time to reach maximum (peak) plasma concentration (Tmax) of tebotelimab and tebotelimab plus margetuximab | At the end of infusion on Study Days 1, 15, 29 and 43 in Cycles 1 and 2 and on Study Day 1 for all subsequent cycles until treatment discontinuation, up to 2 years
  Tmax
Trough plasma concentration (Ctrough) of tebotelimab | Study Days 1, 15, 29, 43 in Cycles 1 and 2 and Day 1 of each subsequent cycle s until treatment discontinuation, up to 2 years
  Ctrough
Total body clearance of the drug from plasma (CL) of tebotelimab | Cycle 1 Day 1 out to Cycle 1 Day 15
  CL
Apparent volume of distribution at steady state (Vss) of tebotelimab | Cycle 1 Day 1 out to Cycle 1 Day 15
  Vss
Terminal half-life (t1/2) of tebotelimab | Cycle 1 Day 1 out to Cycle 1 Day 15
  t1/2
Number of patients with anti-drug antibody | Study Day 1, 15, 29, 57, 85, 113, then every 56 days up to 2 years Tebotelimab plus margetuximab: Day 1, 22, 43, and then every 6 weeks until treatment discontinuation
  immunogenicity
Objective response rate (ORR) | Throughout the study, up to 4 years.
  ORR is the percentage of participants who have a complete response or a partial response to treatment.
Median Duration of response (DoR) | Throughout the study, up to 4 years.
  DoR is defined as the time from the date of initial response (CR or PR) to the date of first documented PD or death from any cause, whichever occurs first. Median DoR is the time when 50% of responders are still in response.
Progression-free survival (PFS) | Throughout the study, up to 4 years.
  PFS is defined as the time from the first dose date to the date of first documented PD or death from any cause, whichever occurs first. Median PFS is the time when 50% of participants remain free of PD or death.
Median Overall survival (OS) | Throughout the study, up to 4 years.
  OS is defined as the time from the first dose date to the date of death from any cause. Median OS is the time when 50% of participants are still alive.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ward, MD, Study Director — MacroGenics
Locations (39):
- United States (15):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital and Dana-Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Stephenson Cancer Center, The University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Australia (4):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Austin Health Melbourne, Heidelberg, Victoria
- Bulgaria (3):
  - "Complex Oncology Center - Burgas" EOOD, Burgas
  - "Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda" EAD, Sofia, Sofia
  - Multiprofile Hospital for Active Treatment "Serdika" EOOD, Sofia, Sofia
- Prince of Wales Hospital, Shatin, Hong Kong
- Poland (4):
  - Pratia MCM Kraków, Krakow, Lesser Poland Voivodeship
  - BioVirtus Research Site Sp. Z o.o. / Biovirtus Centrum Medyczne, Józefów, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Med-Polonia Sp. z o.o., Poznan
- Spain (3):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Hospital Ruber Internacional, Madrid
  - START Madrid-CIOCC, Hospital HM Sanchinarro, Madrid
- Thailand (3):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Songklanagarind Hospital, Songkhla
- Ukraine (6):
  - Communal Nonprofit Enterprise "Cherkassy Regional Oncology Dispensary" of Cherkassy Regional Council, Cherkassy, Cherkasy Oblast
  - Communal Nonprofit Enterprise Podillia Regional Center of Oncology of Vinnytsia Regional Council, Vinnytsia, Vinnytsa Region
  - Communal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, Dnipro
  - Communal Nonprofit Enterprise "Prykarpatsky Clinical Oncological Centre of Ivano-Frankivska Regional Council", Ivano-Frankivsk
  - Municipal Non-Profit Enterprise of Sumy Regional Council "Sumy Regional Clinical Oncology Dispensary", Sumy
  - Communal Nonprofit Enterprise "Central City Clinical Hospital of Uzhhorod City Council", City Oncology Center, State Higher Educational Institution <<Uzhhorod National University>>, Uzhhorod

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luke JJ, Patel MR, Blumenschein GR, Hamilton E, Chmielowski B, Ulahannan SV, Connolly RM, Santa-Maria CA, Wang J, Bahadur SW, Weickhardt A, Asch AS, Mallesara G, Clingan P, Dlugosz-Danecka M, Tomaszewska-Kiecana M, Pylypenko H, Hamad N, Kindler HL, Sumrow BJ, Kaminker P, Chen FZ, Zhang X, Shah K, Smith DH, De Costa A, Li J, Li H, Sun J, Moore PA. The PD-1- and LAG-3-targeting bispecific molecule tebotelimab in solid tumors and hematologic cancers: a phase 1 trial. Nat Med. 2023 Nov;29(11):2814-2824. doi: 10.1038/s41591-023-02593-0. Epub 2023 Oct 19. PMID 37857711